CLINICAL TRIAL: NCT01165450
Title: Phase 2, Randomized, Double-masked, Vehicle-controlled, Dose-escalation Study Evaluating Efficacy/Safety of Nexagon in Subjects With Persistent Corneal Epithelial Defects (PED) Resulting From Corneal Epithelial Debridement During Diabetic Vitrectomy Surgery, Herpes Simples Virus (HSV) Keratitis, Herpes Zoster Virus (HZV) Keratitis, Corneal Burns, Post-photorefractive Keratectomy (Post-PRK), or Post-corneal Transplant Surgery.
Brief Title: Efficacy and Safety Study of Nexagon for Persistent Corneal Epithelial Defects
Acronym: NTX-PED-001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug manufacturer could not supply study drug.
Sponsor: University of California, San Francisco (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nex001; 1R01FD003708-01A1 (FDA)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Persistent Corneal Epithelial Defects
Keywords: persistent epithelial defect; cornea
MeSH Terms: conditions — Corneal Diseases | interventions — Poloxamer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nexagon (Active Comparator): There will be 3 groups of patients with persistent epithelial defects, treated in a dose-escalation fashion from 1µg to 3µg to 10 µg. Each group will consist of 18 patients randomized to Nexagon and 6 patients randomized to placebo only.
  Interventions: Drug: Nexagon
- Vehicle only (Placebo Comparator): There will be 3 groups of patients with persistent epithelial defects, treated in a dose-escalation fashion from 1µg to 3µg to 10 µg. Each group will consist of 18 patients randomized to Nexagon and 6 patients randomized to placebo only.
  Interventions: Drug: Vehicle only

INTERVENTIONS:
Drug: Nexagon — There will be 3 groups of patients with persistent epithelial defects, treated in a dose-escalation fashion from 1µg to 3µg to 10 µg. Each group will consist of 18 patients randomized to Nexagon and 6 patients randomized to placebo only.
  Other Names: Active Ingredient: CODA001; IND: 104593; Vehicle: Poloxamer 407
  Arms: Nexagon
Drug: Vehicle only — There will be 3 groups of patients with persistent epithelial defects, treated in a dose-escalation fashion from 1µg to 3µg to 10 µg. Each group will consist of 18 patients randomized to Nexagon and 6 patients randomized to placebo only.
  Other Names: Poloxamer 407
  Arms: Vehicle only

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nexagon® in subjects with persistent corneal epithelial defects (PED) resulting from corneal epithelial debridement during diabetic vitrectomy surgery, HSV keratitis, HZV keratitis, corneal burns, post-PRK, or post-corneal transplant surgery.

DETAILED DESCRIPTION:
The purpose of this prospective, randomized, double-masked, vehicle-controlled, dose-escalation study is to evaluate the efficacy and safety of Nexagon® in subjects with persistent corneal epithelial defects (PED) resulting from corneal epithelial debridement during diabetic vitrectomy surgery, HSV keratitis, HZV keratitis, corneal burns, post-PRK, or post-corneal transplant surgery. In general, traditional therapy of PED consists of aggressive lubrication with preservative-free artificial tears and ointments, the use of bandage soft contact lenses, pressure patching, punctal plugging, and the surgical closure of the eyelids. Unfortunately, the success rates with these conventional treatment modalities are varied, and overall, disappointingly low. As such, much research is currently being directed at finding better treatments for PED. Nexagon® is a novel therapeutic agent that has been shown to be effective in treating skin lesions, and it has been shown in animal studies and in preliminary human studies to be safe and efficacious in treating PED.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years and over.
* Female subjects must be a) postmenopausal, b) surgically sterilized, c) practicing abstinence, or d) using a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide for the duration of the study.
* Subjects who are able to attend all follow-up visits and who are able to comply with all study procedures.
* Subjects who are willing and able to give written informed consent to take part in the study.
* Subjects with a PED, defined as follows: "a corneal epithelial defect persisting for at least 14 days and not longer than 28 days."
* In the Investigator's opinion, the defect is persistent i.e., the defect has not shown improvement despite conventional treatment such as tear supplements and bandage contact lenses.
* The original defect to the cornea must have resulted from corneal epithelial debridement during diabetic vitrectomy surgery, HSV keratitis, HZV keratitis, corneal burns, post-PRK, or post-corneal transplant surgery.

Exclusion Criteria:

* Use of concomitant ocular medications in the screening period that are not specified in standardized PED treatment regimen
* Likely to require the use of concomitant ocular medications that are not specified in the standardized PED treatment regime during the study follow-up period
* Decrease or increase in the PED by more than 50% during the screening period.
* Have an active eyelid or ocular infectious process of any sort, in the opinion of the Investigator.
* Subjects with corneal perforation or impending corneal perforation.
* Subjects with severe eyelid abnormalities contributory to the persistence of the PED.
* Subjects with bilateral PED, if the smaller PED has a longest diameter of > 2 mm. (Note: if bilateral PED is present and the smaller PED is < 2 mm, the subject is eligible. In this situation only the eye with the larger PED should be entered into the study).
* Female subjects who are pregnant or breastfeeding. Female subjects who are neither postmenopausal nor surgically sterile require a negative urine pregnancy test on Day 0 (plus or minus 1 day) visit.
* Subjects who have a history of AIDS or HIV.
* Subjects with any other condition which, in the Investigator's opinion, would exclude the subject from participating.
* Treatment with systemic corticosteroids (equivalent to > 10 mg/day of prednisone) or immunosuppressive or chemotherapeutic agents within 7 days prior to Day 0 (plus or minus 1 day) visit, or likely to receive one of these therapies during study participation
* Subjects who have participated in a clinical trial within 30 days prior to Day 0 (plus or minus 1 day) visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bennie H Jeng, MD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Qiu C, Coutinho P, Frank S, Franke S, Law LY, Martin P, Green CR, Becker DL. Targeting connexin43 expression accelerates the rate of wound repair. Curr Biol. 2003 Sep 30;13(19):1697-703. doi: 10.1016/j.cub.2003.09.007. PMID 14521835
- [Background] Lin JH, Weigel H, Cotrina ML, Liu S, Bueno E, Hansen AJ, Hansen TW, Goldman S, Nedergaard M. Gap-junction-mediated propagation and amplification of cell injury. Nat Neurosci. 1998 Oct;1(6):494-500. doi: 10.1038/2210. PMID 10196547

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients were enrolled but only 2 randomized. The third patient was withdrawn from the trial before randomization because we were notified that the study drug had expired and was no longer available.
Groups:
- Overall Study: We enrolled three patients and randomized and treated two patients in the first cohort. On October 24, 2012 we were notified by David Eisenbud, MD (Chief Medical Officer, CoDa Therapeutics, Inc) that our supply of low dose study drug was expired and no more would be produced by the drug manufacturer.
Period: Overall Study
Arm/Group | Overall Study
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2 participants were randomized and participated in the study before its premature closure for lack of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Healing of the Corneal Epithelial Defect at Day 14 ± 1 in the Study Eye
Description: Primary efficacy measure: To determine whether topical treatment of persistent epithelial defects with Nexagon preparations yields greater healing at Day 14 ± 1, compared to vehicle alone, in individuals having had diabetic vitrectomy. Healing will be determined by comparing pseudo-area (as measured by Investigator, or designated ophthalmologist) at baseline (taken just prior to the first treatment) and Day 14 ± 1. Pseudo-area is defined by the longest diameter of the lesion multiplied by the longest perpendicular to this longest diameter.
Time Frame: 14 ± 1 days
Population: The study was terminated prematurely, data were never analyzed; PI has left the institution and data are no longer available.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence of Adverse Events Following Application of the Investigational Product in All Subjects
Description: Primary safety measure: To determine incidence of adverse events by recording their occurrence at each study visit through Day 28 ± 2. Analysis of safety data will be performed prior to each dose-escalation. If greater than 2 serious adverse events are found that are causally related to the investigational product, the study will be halted.
Time Frame: 28 ± 2 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Complete Re-epithelialization of the Study Eye
Description: Resolution of epithelial defect is defined as the largest diameter of the epithelial defect being less than 0.5 mm, as it is difficult to distinguish a smaller defect from the small amount of fluorescing staining seen in a healed defect. Time of complete re-epithelialization will be defined as the midpoint between the last observed date with an epithelial defect and the date of the first visit with no epithelial defect, up to Day 28 ± 2.
Time Frame: 28 ± 2 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Complete Healing of the Corneal Epithelial Defect at Day 14 ± 1 in the Study Eye
Description: To determine binary indicator of whether or not healing has occurred at 14 ± 1 days, defined as the largest diameter of the epithelial defect being smaller than 0.5 mm as determined by slit lamp examination with fluorescein staining.
Time Frame: 14 ± 1 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in the Rate of Re-epithelialization of the Study Eye
Description: To determine the change in the rate of re-epithelialization of the study eye from the screening run-in period to the treatment period, if applicable.
  Time Frame: Screening period is defined as Day -7 to Day 0 ± 1. Treatment period is defined as Day 0 ± 1 through time of complete re-epithelialization. Time of complete re-epithelialization is defined as the midpoint between the last observed date with an epithelial defect and the date of the first visit with no epithelial defect, up to Day 28 ± 2.
Time Frame: 35 ± 2 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Persistence of Complete Corneal Re-epithelialization in the Study Eye
Description: To determine whether or not complete corneal re-epithelialization was persistent, as determined by whether the healed epithelium remains intact after complete re-epithelialization is confirmed in the study eye. The measurement will be made at Day 28 ± 2.
Time Frame: 28 ± 2 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

7. Secondary Outcome: Percent Reduction of Corneal Epithelial Defect at Day 28 ± 2 in the Study Eye
Description: To compare, in each of the two patient populations, the percent reduction in epithelial defect size at Day 28 ± 2 compared to baseline, as measured by slit lamp examination with fluorescein staining. Epithelial defect size determined by pseudo-area, defined by the longest diameter of the lesion multiplied by the longest perpendicular to this longest diameter.
Time Frame: 28 ± 2 days
Population: as for outcome 1
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to discontinued supply of study drug, and data were never analyzed; PI has left the institution and data are no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes